CLINICAL TRIAL: NCT02193243
Title: The Diagnostic Value of Six-Minute Walk Test in Grown-Up Patients With Congenital Heart Disease (GUCH)
Brief Title: Value of 6-minute Walk Test in Grown Ups With Congenital Heart Defects (GUCH)
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Disease and Vascular Medicine, Heinrich-Heine University, Duesseldorf
Other Study IDs: Six-Minute Walk Test
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Six Minute Walk Test; Exercise Testing; Peak oxygen uptake
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The six-minute walk test is an established submaximal exercise test. Its role in examination of grown-up patients with congenital heart disease (GUCH) is not studied so far. Objective of this study was a comparison of the 6MWT with other established parameters of functional capacity, in grown-up patients with GUCH.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart defect
* > 18 years

Exclusion Criteria:

* mental or physical incapability of exercise testing
* non-cardiac limitations of physical capacity, as e.g. orthopedic diseases or febrile infections
* severe psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with Congenital Heart Disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Ranges of six-minute walk distance (6MWD) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eva S Kehmeier, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Heinrich Heine University Div. of Cardiology, Pulmonary Disease and Vasculae Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Kehmeier ES, Sommer MH, Galonska A, Zeus T, Verde P, Kelm M. Diagnostic value of the six-minute walk test (6MWT) in grown-up congenital heart disease (GUCH): Comparison with clinical status and functional exercise capacity. Int J Cardiol. 2016 Jan 15;203:90-7. doi: 10.1016/j.ijcard.2015.10.074. Epub 2015 Oct 22. PMID 26498869